CLINICAL TRIAL: NCT04657679
Title: evaLuation of Variations pharmacokinEtics and phArmacogeNOmics of Ribociclib in rAce-based Cohorts: The LEANORA Study
Brief Title: Pharmacokinetics and Pharmacogenomics of Ribociclib in Race-based Cohorts
Acronym: LEANORA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sufficient accrual into the African American/Black patient cohort and insufficient accrual into the NHW patient cohort.
Sponsor: Georgetown University (Other)
Collaborators: Medstar Health Research Institute (Other); Breast Cancer Research Foundation (Other); Georgetown-Howard Universities Center for Clinical and Translational Science (GHUCCTS) (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00003100
Record Dates: First submitted 2020-11-20; First posted 2020-12-08 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: HR-positive/HER2-negative metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- African American/Black (Active Comparator): Subject who self identify as African American or Black with metastatic HR+/HER2- advanced breast cancer (estimate 3 participants who are CYP3A5 poor metabolizers and approximately 15 participants who are CYP3A5 intermediate or normal metabolizers)
  Interventions: Drug: Ribociclib
- Non-Hispanic White (Active Comparator): Subjects who self-identify as non-Hispanic White with metastatic HR+/HER2- advanced breast cancer (estimate 3 participants who are CYP3A5 poor metabolizers and approximately 15 participants who are CYP3A5 intermediate or normal metabolizers)
  Interventions: Drug: Ribociclib

INTERVENTIONS:
Drug: Ribociclib — Patients will receive ribociclib 600 mg oral (PO) daily for 21 consecutive days of 28-day cycles and endocrine therapy with either letrozole or fulvestrant. Fulvestrant 500 mg intramuscular (IM) will be administered on days 1, 15, 29 of cycle one, and then monthly. Letrozole 2.5 mg oral daily continuously. If premenopausal women have not undergone bilateral salpingo- oophorectomy, they will receive a luteinizing hormone-releasing hormone (LHRH) agonist (e.g., goserelin leuprolide) for ovarian suppression in combination with fulvestrant or letrozole and ribociclib.
  Other Names: KISQALI

SUMMARY:
The aim is to determine the pharmacological and biochemical association between ribociclib exposure and CYP3A variants in African American/Blacks and Non-Hispanic White patients. The investigators hypothesize that patients treated with ribociclib who are CYP3A5 poor metabolizers may be exposed to higher levels of ribociclib than CYP3A5 intermediate or normal metabolizers. The findings could allow clinicians to tailor treatments to maintain therapeutic doses while limiting toxicities.

DETAILED DESCRIPTION:
This prospective, multicenter, cohort study will assess ribociclib (600 mg PO daily) pharmacokinetics and pharmacogenomics in female patients with HR+/HER2- metastatic breast cancer. This design will be used for two independent, race-based cohorts: 18 African American/Black patients and 18 Non-Hispanic White patients. Women are eligible if they are older than 18, have HR+/HER2- mBC and are candidates for treatment with a CDK 4/6 inhibitor and endocrine therapy. Patients are ineligible if currently prescribed a medication that inhibits or induces the CYP3A isoenzymes, have baseline electrocardiogram abnormalities, or are otherwise considered to be ineligible for ribociclib. Participants will provide serial blood samples during the first cycle (collected immediately prior to the ribociclib dose, and 0.5hr ± 5min, 1hr ± 5min, 2hr ± 15min, 4hr ± 15min, 6hr ± 15min after the daily dose of ribociclib). Plasma samples will be analyzed via mass spectrometry to characterize the pharmacokinetics (e.g., AUC0-24, Cmax). Pharmacogenetic testing will be performed using the PharmacoScanTM microarray, which tests 4,627 markers in 1,191 genes, including variants in CYP3A4 and CYP3A5.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to any screening procedures.
* Female ≥18 years old at the time of informed consent
* Those who self-identify as African American or Black are eligible for that respective cohort
* Those who self-identify as non-Hispanic White are eligible for that respective cohort
* Postmenopausal or premenopausal. Patient has a known menopausal status at the time of the informed consent form signature. The patient is considered postmenopausal if: i) she has had prior bilateral oophorectomy; ii) is age ≥ 60 years; iii) is age <60 years and has had amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression) and follicle-stimulating hormone (FSH) and estradiol in the postmenopausal range per local normal ranges. All other patients who do not meet the criteria for postmenopausal status are considered premenopausal and will receive goserelin or leuprolide for ovarian suppression
* Each race-based cohort has a predetermined number of patients with each CYP3A5 phenotype per the sample size calculation (section 9.1). Patients will be screen for CYP3A5: - African American or Black (At least 3 participants who are CYP3A5 poor metabolizers, No more than 15 participants who are CYP3A5 intermediate or normal metabolizers); - Non-Hispanic White (At least 3 participants who are CYP3A5 intermediate or normal metabolizers, No more than 15 participants who are CYP3A5 poor metabolizers)
* Patient has advanced (loco-regionally recurrent or metastatic) breast cancer not amenable to curative therapy
* Treated, stable and asymptomatic brain metastases are permitted
* ECOG performance status 0-3
* Documentation of estrogen receptor (ER) positive and/or progesterone receptor (PR) positive tumor (≥1% positive stained cells) based on most recent tumor biopsy (discuss with the Principal Investigator if results in different biopsies are discordant in terms of hormone receptor positivity) utilizing an assay consistent with local standards.
* Documented HER2-negative tumor based on local testing on most recent tumor biopsy: HER2-negative tumor is determined as immunohistochemistry score 0/1+ or negative by in situ hybridization (FISH/CISH/SISH) defined by current ASCO/CAP (American Society of Clinical Oncology/College of American Pathologists) guidelines. Patients with equivocal HER2 in situ hybridization results according to current ASCO/CAP guidelines are eligible, as long as they have not received and are not scheduled to receive anti-HER2 treatment.
* Must be capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by the IRB, prior to the initiation of any screening or study-specific procedures.
* Patient must be able to swallow ribociclib tablets.
* Patient must be able to communicate with the investigator and comply with the requirements of the study procedures.
* Patient has adequate bone marrow and organ function as defined by the following laboratory values:

  1. Absolute neutrophil count (ANC) ≥ 1,200/mm; Patients must be able to meet the criteria without receipt of colony stimulating factors within 2 weeks before obtaining sample
  2. Platelets ≥ 100,000/mm3; Patients must be able to meet the criteria without receipt of transfusion within 2 weeks before obtaining sample
  3. Hemoglobin ≥ 8 g/dL; Patients must be able to meet the criteria without receipt of transfusion within 2 weeks before obtaining sample
  4. Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73m2 according to the CKD EPI equation
  5. Total bilirubin < ULN except for patients with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN.
  6. Aspartate transaminase (AST) < 2.5 × ULN, except for patients with liver metastases, who are only included if the AST is <5 × ULN.
  7. Alanine transaminase (ALT) < 2.5 × ULN, except for patients with liver metastases, who are only included if the ALT is < 5 × ULN.
  8. Alkaline phosphatase ≤2.5 x ULN (≤5.0 x ULN if bone metastases present)
* Patient must have the following laboratory values within normal limits or corrected to within normal limits with supplements, or are not clinically significant per the Investigator

  1. Sodium
  2. Potassium
  3. Calcium
* The following tests are not necessary. However, if results are available, values should be as follows:

  * INR ≤ 1.5 (unless the patient is receiving anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to the first dose of study drug).
  * Magnesium within normal limits or corrected to within normal limits with supplements, or is not clinically significant per the Investigator.
* Standard 12-lead electrocardiogram values defined as (obtained from baseline electrocardiogram):

  1. QTc interval at screening < 450 ms (using Fridericia's correction)
  2. Mean resting heart rate >= 50 bpm (determined from the electrocardiogram)

Exclusion Criteria:

* Patient with symptomatic visceral disease or any disease burden that makes the patient ineligible for endocrine therapy per the investigator's judgment.
* Patient currently prescribed a CDK4/6 inhibitor (e.g., ribociclib, abemaciclib, or palbociclib).
* Patients with central nervous system (CNS) symptomatic or untreated metastases
* History of liver transplant or allogeneic bone marrow transplantation
* Patient with a known hypersensitivity to any of the excipients of ribociclib (e.g. ribociclib tablets coating contains soya lecithin, and therefore should not be taken by patients who are allergic to peanuts or soya) or of fulvestrant.
* Patient is concurrently using other anti-cancer therapy besides those in the study protocol (e.g., letrozole, fulvestrant, goserelin, leuprolide). Any other prior neo-/adjuvant anti-cancer therapy must be stopped at least 5 half-lives or 7 days, whichever is longer, before the date of ribociclib initiation.
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major toxicities
* Patient has not recovered from acute clinical and laboratory toxicities related to prior anticancer therapies to NCI CTCAE v5.0 grade ≤ 1 (except for alopecia, neuropathy, and amenorrhea or other toxicities not considered a safety risk for the patient at investigator's discretion).
* Patient has received extended-field radiotherapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to ribociclib initiation and has not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).
* Patient has a concurrent malignancy, with the exception of adequately treated basal or squamous cell skin carcinoma, stage 1 melanoma, or curatively resected cervical carcinoma in situ. Patients may still enroll with a concurrent malignancy after receiving approval from the study PI.
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drug (e.g., uncontrolled ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patient has any other concurrent severe and/or uncontrolled medical condition that would in the investigator's judgment, cause unacceptable safety risks to the patient, contraindicate patient participation in the clinical study, or compromise compliance with the protocol.
* Patient has clinically significant, uncontrolled heart disease or who are at significant risk of developing QT prolongation, including any of the following:

  1. Documented myocardial infarction (MI), angina pectoris, coronary artery intervention, or pericarditis within 6 months prior to study entry
  2. Documented cardiomyopathy, congestive heart failure, valvular heart disease, congenital heart disease, or prior cardiac surgery
  3. Left Ventricular Ejection Fraction (LVEF) < 50% (testing is not mandatory)
  4. Personal diagnosis of long QT syndrome, cardiac channelopathies, family history of idiopathic sudden death, congenital long QT syndrome or channelopathies
  5. Personal risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia, hypomagnesemia, or need for concomitant medications with a known risk to prolong the QT interval and/or known to cause TdP that cannot be discontinued or replaced by safe alternative medication (e.g. within 5 half-lives or 7 days prior to starting study drug, whichever is longer)
  6. Clinically significant cardiac arrhythmias or conduction abnormalities, including, but not limited to ventricular tachycardia, atrial tachyarrhythmia, left bundle branch block, right bundle branch block, QRS prolongation (greater than 120 ms), intraventricular conduction delay, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block)
  7. Uncontrolled hypertension
  8. Inability to determine the QTc interval
* Patient is currently receiving any of the following substances and cannot be discontinued 7 days prior to Cycle 1 Day 1:

  1. Concomitant medications, herbal supplements, and/or fruits that are strong inducers or inhibitors of CYP3A4/5.
  2. Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
  3. Chronic dosing of corticosteroids such as dexamethasone and prednisone is known to lead to induction of CYP3A enzymes, thereby potentially reducing ribociclib drug exposure to sub-therapeutic levels. Systemic corticosteroid treatment should not be given during the study treatment with ribociclib, except for:

     * Topical applications (e.g. for rash), inhaled sprays (e.g. for obstructive airways diseases), eye drops or local injections (e.g. intra-articular)
     * A short duration (< 5 days) of systemic corticosteroids ≤ to the anti-inflammatory potency of 4 mg dexamethasone (e.g. for chronic obstructive pulmonary disease or as an antiemetic).
     * Medications that prolong the QTc interval.
* Inability to comply with study requirements.
* Psychiatric illness or social situation that would limit compliance with study requirements.
* Patients with clinically significant liver disease, including active viral or other known hepatitis, current alcohol abuse, or cirrhosis.
* Known active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg]) or known active hepatitis C (defined as a positive test for hepatitis C viral load by polymerase chain reaction [PCR]).

  * Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible.
  * Patients with positive hepatitis C antibody AND negative quantitative hepatitis C by PCR AND no clinical/laboratory evidence of cirrhosis are eligible. Patients who have completed curative therapy for HCV are eligible if they meet all other parameters for enrollment.
  * Patients are not required to undergo testing for HBV or HCV for enrollment
* Known uncontrolled HIV infection defined as any of the following 3 criteria:

  * CD4 counts ≤ 350 cells/μL; or
  * Serum HIV viral load ≥ 400 copies/mL; or
  * Have been taking an antiretroviral regimen for < 4 weeks prior to treatment with study drugs if anti-retroviral therapy is deemed necessary or appropriate by the investigator.
  * Patients are not required to undergo testing for HIV for enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Swain, MD, Principal Investigator — Georgetown University
Locations (3):
- United States (3):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Tufts Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | African American/Black | Non-Hispanic White
Started | 17 | 4
Completed | 14 | 3
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | African American/Black | Non-Hispanic White | Total
Number analyzed (Participants) | 17 | 4 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 1 | 12
  >=65 years | 6 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 4 | 21
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 4 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 0 | 17
  White | 0 | 4 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
CYP3A5 phenotype [Count of Participants; unit: Participants]
  IM/NM: intermediate metabolizers/normal metabolizers | 9 | 0 | 9
  PM: poor metabolizers | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Ribociclib Area-under-the-curve (AUC)
Description: Compare the exposure (i.e., AUC) of ribociclib at steady-state between CYP3A5 poor metabolizers (PM) and CYP3A5 intermediate or normal metabolizers (IM/NM) in each independent race-based cohort of women with advance breast cancer
Time Frame: On day 8-16 of cycle 1 (each cycle is 28 days)
Population: One subject in the Non-Hispanic white arm was excluded to prohibited medication. All Non-Hispanic white participants were in the CYP3A5 Poor Metabolizers (PM) group.
Measure: Median (Inter-Quartile Range); unit: hr*ng/mL
Arm/Group | African American/Black | Non-Hispanic White
Number analyzed (Participants) | 14 | 3
hr*ng/mL
  CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  CYP3A5 IM/NM | 43546 [35298 to 46647] |
  CYP3A5 PM: number analyzed (Participants) | 7 | 3
  CYP3A5 PM | 39230 [18745 to 57566] | 33230 [17142 to 39492]

2. Secondary Outcome: Ribociclib Pharmacokinetic Properties - Maximum Concentration (Cmax)
Description: Maximum concentration (Cmax) at steady state between different CYP3A5 phenotypes
Time Frame: On day 8-16 of cycle 1 (each cycle is 28 days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | African American/Black | Non-Hispanic White
Number analyzed (Participants) | 14 | 3
ng/mL
  Cmax CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  Cmax CYP3A5 IM/NM | 3140 [1980 to 3540] |
  Cmax CYP3A5 PM: number analyzed (Participants) | 7 | 3
  Cmax CYP3A5 PM | 3020 [1300 to 3470] | 2300 [2220 to 2640]

3. Secondary Outcome: Ribociclib Pharmacokinetic Properties - the Time to Reach Cmax (Tmax)
Description: the time to reach Cmax (Tmax) at steady state between different CYP3A5 phenotypes
Time Frame: On day 8-16 of cycle 1 (each cycle is 28 days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | African American/Black | Non-Hispanic White
Number analyzed (Participants) | 14 | 3
hour
  CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  CYP3A5 IM/NM | 2.0 [2.0 to 4.0] |
  CYP3A5 PM: number analyzed (Participants) | 7 | 3
  CYP3A5 PM | 3.8 [2.0 to 5.9] | 0.97 [0.58 to 4.1]

4. Secondary Outcome: Ribociclib Pharmacokinetic Properties - Clearance
Description: clearance at steady state between different CYP3A5 phenotypes
Time Frame: On day 8-16 of cycle 1 (each cycle is 28 days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: liter/hour
Arm/Group | African American/Black | Non-Hispanic White
Number analyzed (Participants) | 14 | 3
liter/hour
  CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  CYP3A5 IM/NM | 13.78 [12.86 to 17.00] |
  CYP3A5 PM: number analyzed (Participants) | 7 | 3
  CYP3A5 PM | 15.29 [10.42 to 32.00] | 18.06 [15.19 to 35.00]

5. Secondary Outcome: Ribociclib Pharmacokinetic Properties - Volume of Distribution(vd)
Description: Volume of distribution(vd) at steady state between different CYP3A5 phenotypes
Time Frame: days 8-16 of cycle 1 (28 day cycle)
Population: One subject in the Non-Hispanic white arm was excluded due to prohibited medication.
Measure: Median (Inter-Quartile Range); unit: Liters
Arm/Group | African American/Black | Non-Hispanic White
Number analyzed (Participants) | 14 | 3
Liters
  CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  CYP3A5 IM/NM | 413.88 [370.75 to 520.77] |
  CYP3A5 PM: number analyzed (Participants) | 7 | 3
  CYP3A5 PM | 465.33 [319.72 to 813.19] | 455.90 [438.76 to 954.99]

6. Secondary Outcome: Ribociclib Pharmacokinetic Properties - Elimination Half-life
Description: Elimination half-life (t1/2) at steady state between different CYP3A5 phenotypes
Time Frame: On day 8-16 of cycle 1 (each cycle is 28 days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | African American/Black | Non-Hispanic White
Number analyzed (Participants) | 14 | 3
hour
  CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  CYP3A5 IM/NM | 21.24 [20.61 to 25.12] |
  CYP3A5 PM: number analyzed (Participants) | 7 | 3
  CYP3A5 PM | 21.26 [21.09 to 22.70] | 18.91 [17.50 to 20.02]

7. Secondary Outcome: Change in QTc Interval
Description: Change in QTc interval between 1) baseline and between days 8-16 of cycle 1 (midcycle), and 2) baseline and scheduled visit prior to initiation of cycle 2 (C2), between different CYP3A5 phenotypes.
Time Frame: Baseline, day 8-16 of cycle 1 and prior to cycle 2 (each cycle is 28 days)
Population: One subject in the Non-Hispanic white arm was excluded to prohibited medication.
Measure: Median (Inter-Quartile Range); unit: Change in ms
Arm/Group | African American/Black | Non-Hispanic White
Number analyzed (Participants) | 14 | 3
Change in ms
  MidCycle -CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  MidCycle -CYP3A5 IM/NM | 19 [0 to 37] |
  MidCycle- CYP3A5 PM: number analyzed (Participants) | 7 | 3
  MidCycle- CYP3A5 PM | -7 [-11 to 16] | 23 [23 to 36]
  Prior to C2- CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  Prior to C2- CYP3A5 IM/NM | 11 [-26 to 29] |
  Prior to C2- CYP3A5 PM: number analyzed (Participants) | 7 | 3
  Prior to C2- CYP3A5 PM | -4 [-17 to 5] | 31 [23 to 40]

8. Secondary Outcome: Laboratory Abnormalities - Neutropenia
Description: Occurrence of neutropenia
Time Frame: from baseilne through prior to cycle 2 (each cycle is 28 days)
Population: One subject in the Non-Hispanic white arm was excluded to prohibited medication.
Measure: Count of Participants; unit: Participants
Arm/Group | African American/Black | Non-Hispanic White
Number analyzed (Participants) | 14 | 3
Participants
  CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  CYP3A5 IM/NM | 0 |
  CYP3A5 PM: number analyzed (Participants) | 7 | 3
  CYP3A5 PM | 3 | 1

9. Secondary Outcome: Laboratory Abnormalities - Aspartate Aminotransferase (AST)
Description: Occurrence of Laboratory abnormalities: AST
Time Frame: From Baseline through prior to cycle 2 (each cycle is 28 days)
Population: One subject in the Non-Hispanic white arm was excluded to prohibited medication.
Measure: Count of Participants; unit: Participants
Arm/Group | African American/Black | Non-Hispanic White
Number analyzed (Participants) | 14 | 3
Participants
  CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  CYP3A5 IM/NM | 0 |
  CYP3A5 PM: number analyzed (Participants) | 7 | 3
  CYP3A5 PM | 1 | 0

10. Secondary Outcome: Laboratory Abnormalities -Alanine Aminotransferase (ALT)
Description: Occurrence of Laboratory abnormalities: ALT between between different CYP3A5 phenotypes.
Time Frame: From Baseline to prior to cycle 2 (each cycle is 28 days)
Population: One subject in the Non-Hispanic white arm was excluded to prohibited medication.
Measure: Count of Participants; unit: Participants
Arm/Group | African American/Black | Non-Hispanic White
Number analyzed (Participants) | 14 | 3
Participants
  CYP3A5 IM/NM: number analyzed (Participants) | 7 | 0
  CYP3A5 IM/NM | 1 |
  CYP3A5 PM: number analyzed (Participants) | 7 | 3
  CYP3A5 PM | 1 | 0

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | African American/Black | Non-Hispanic White
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/3
Other Adverse Events (participants affected / at risk) | 14/14 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | African American/Black (N=14) | Non-Hispanic White (N=3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | African American/Black (N=14) | Non-Hispanic White (N=3)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 4 (6) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) — mouth sores
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (7) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) — COVID-19
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
QTc Prolongation (Cardiac disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT04657679/Prot_SAP_000.pdf